CLINICAL TRIAL: NCT03117725
Title: Comparison of IVF Outcome and Endometrium Effect in Infertility Patients Between Diminished and Normal Ovarian Reserve After Melatonin Administration.
Brief Title: Melatonin Study Between Diminished and Normal Responder in IVF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Bundang CHA Hospital (Other)
Responsible Party: Principal Investigator, Dong Hee Choi, M.D, Ph.D, Bundang CHA Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2016-07-013-008
Record Dates: First submitted 2017-04-04; First posted 2017-04-18 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Infertility, Female
Keywords: oxidative stress; antioxidants; diminished ovarian reserve
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- melatonin administration group (Experimental): Total 50 patients are to be randomized into this group, 25 of which are poor responder and the others are normal responders. After randomization, participants are to under go melatonin administration intervention from the time of controlled ovarian hyperstimulation(COH) to the date of oocyte retrieval. If pregnancy is not confirmed in the first cycle, all subjects are to enter the second cycle after 1-2 months of recovery period.
  For the second cycle, the procedure will be repeated same as the first cycle with doubling of the drug dosage . It should also be administered for 2 weeks until the date of oocyte retrieval.
  Interventions: Drug: Melatonin adminstration
- placebo comparator (Placebo Comparator): Total 50 patients are to be randomized into this group, 25 of which are poor responder and the others are normal responders. Participants for placebo comparator are advised to take the drug (placebo) from the time of COH to the date of oocyte retrieval. If pregnancy is not confirmed in the first cycle, all subjects are to enter the second cycle after 1-2 months of recovery period.
  For the second cycle, the procedure will be repeated same as the first cycle with doubling of the drug dosage . It should also be administered for 2 weeks until the date of oocyte retrieval.
  Interventions: Drug: placebo administration

INTERVENTIONS:
Drug: Melatonin adminstration — The drug, melatonin will be taken every night from the time of COH to the date of oocyte retrieval. The method of administration is as follows: Melatonin 2mg once a day, 1 to 2 hours before bedtime for about 2 weeks until the date of oocyte retrieval.
  Arms: melatonin administration group
Drug: placebo administration — the drug, placebo pill will be taken every night from the time of COH to the date of oocyte retrieval. The method of administration is as follows: placebo pill once a day, 1 to 2 hours before bedtime for about 2 weeks until the date of oocyte retrieval.
  Arms: placebo comparator

SUMMARY:
Poor sleep quality may lead to increase in oxidative stress and free radicals which in turn may decrease the reproductive function. Many researchers have already proven improvement on reproductive function after antioxidant (melatonin) administration. The investigators wish to study the relationship between unexplained, young poor ovarian responder and oxidative stress.

DETAILED DESCRIPTION:
Poor sleep quality may lead to increase in oxidative stress and free radicals which in turn may decrease the reproductive function. Many researchers have already proven improvement on reproductive function after antioxidant (melatonin) administration. The investigators wish to study the relationship between unexplained, young poor ovarian responder and oxidative stress.

This is an randomized controlled trial to evaluate the effect of melatonin to improve the quality of sleep and reduce the oxidative stress. 100 patients will be randomized in to two groups, the one with melatonin administration for 2 weeks and the other with placebo administration. Each group will be composed of 2 sub groups, poor responders and normal responders.

Then the serum and the follicular fluid will be collected at the time of oocyte retrieval and melatonin concentration oxidative stress marker will be measured.

ELIGIBILITY:
Inclusion Criteria:

1. Infertility patients visiting Bundang CHA hospital between the age of 20 to 40.
2. Currently, not being treated for any gynecological or medical diseases.

Exclusion Criteria:

1. Current untreated pelvic pathology (moderate-to-severe endometriosis, submucosal uterine fibroids/polyps assessed by the treating specialist to affect fertility, pelvic inflammatory disease,uterine malformations, and hydrosalpinx.)
2. Currently enrolled in another interventional clinical trial.
3. Concurrent use of other adjuvant therapies (e.g.Chinese herbs, acupuncture).
4. Autoimmune disorders.
5. Undergoing preimplantation genetic diagnosis.
6. Concurrent use of any of the following medications (Fluvoxamine,Cimetidine, Quinolones, Carbamazepine, rifampicin,Zolpidem, zopiclone, and other non-benzodiazepine hypnotic, other CYP1A2 inducers.
7. Genetic disorders regarding galactose intolerance, lactase deficiency, glucose-galactose malabsorption
8. Inability to comply with trial protocol.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-05-12 (Actual); Primary Completion 2019-08-30 (Estimated); Study Completion 2019-10-31 (Estimated)

PRIMARY OUTCOMES:
IVF outcome - oocyte quality | 3 days after oocyte retrieval
  Evaluate oocyte quality on morphological standard as following category- Mature oocyte, Intermediate oocyte, atretic oocyte, post mature oocyte
IVF outcome - embryo quality | 3 to 5 days after oocyte retrieval
  grade the embryos& blastocysts according to the Lucinda Veeck & Gardner
IVF outcome -biochemical pregnancy rate | on day 12~14 after embryo transfer
  serum human chorionic gonadotropin level>10 IU
IVF outcome - clinical pregnancy rate | at 6-8 weeks of gestation
  presence of G-sac in the uterine cavity

SECONDARY OUTCOMES:
acquired oocyte No | 20weeks
  number
fertilization rate | 20weeks
  ratio of no. of fertilized egg/ no of total retrieved eggs
Comparing Pittsburgh sleep quality index | 20weeks
  questionaires to evaluate the participants quality of the sleep. cut off : 13 points This questionaire is to be asked to the participants twice, before and after the administration of the drug
marker(melatonin level, receptor, 8-OHdg) in serum, follicular fluid and endometrium during IVF | 20weeks
  :pg/ml units are used

CONTACTS AND LOCATIONS:
Overall Officials: DONG HEE CHOI, M.D,Ph.D, Principal Investigator — BUNDANGCHA HOSPITAL
Locations (1):
- Bundang CHA medical center, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fernando S, Osianlis T, Vollenhoven B, Wallace E, Rombauts L. A pilot double-blind randomised placebo-controlled dose-response trial assessing the effects of melatonin on infertility treatment (MIART): study protocol. BMJ Open. 2014 Sep 1;4(8):e005986. doi: 10.1136/bmjopen-2014-005986. PMID 25180056
- Available data/document: Study Protocol: 31098 — https://ezdrug.mfds.go.kr